CLINICAL TRIAL: NCT05768529
Title: A Single-arm, Open and Multicenter Phase I/II Clinical Study to Evaluate the Safety and Efficacy of U16 Injection in the Treatment of Refractory/Recurrent B-cell Non-Hodgkin's Lymphoma (r/r B-NHL)
Brief Title: Clinical Study of U16 in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U16-I/II-01
Record Dates: First submitted 2023-02-08; First posted 2023-03-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Non-Hodgkin | interventions — LPAR4 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- U16 (Experimental): Route of administration: Intravenous injection.
  Lymphodepletion conditioning:
  Lymphodepletion will be conducted several days prior to U16 infusion.
  A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  Interventions: Drug: U16

INTERVENTIONS:
Drug: U16 — A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered before U16 treatment.

SUMMARY:
The study is a Phase I/II, single-arm, open-label clinical trial, and its primary objective of phase I and phase II is to evaluate the safety and efficacy of U16 Injection in the treatment of relapsed or refractory NHL,respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to sign the informed consent form and have good compliance;
2. Aged 18-70 years, male or female;
3. CD20-positive B-cell non-Hodgkin's lymphoma with immunohistochemistry(IHC), with the following diagnostic: Diffuse large B cell lymphoma (DLBCL), or Primary mediastinal large B cell lymphoma (PMBCL), or Follicular lymphoma transformed large B cell lymphoma (TFL) , or High grade B cell lymphoma(HGBCL);
4. Previously received≥2nd-line adequate therapy or autologous hematopoietic stem cell transplantation (ASCT), including: a) Received anthracycline-containing drugs and rituximab or other CD20-targeted drugs (except CD20-negative tumors); b) Definition of line: Stable disease (SD) after receiving a first-line therapy for at least 4 cycles or progressive disease (PD), and SD after a second-line therapy for at least 2 cycles or PD; c) For transformed follicular lymphoma (TFL), patients must be treated adequately against FL, and after transformation, must have received at least once the therapy against TFL, and become relapsed or refractory after the last therapy;
5. In relapsed or refractory status at screening: a) Definition of relapse: Remission (including partial remission (PR) or complete remission (CR)) after treatment with at least the standard therapy regimen, and then PD; b)Definition of refractory: i. Non-response to the last therapy: The best response by the last therapy is SD or PD, and the duration is less than 6 months; ii. Relapse or progression (it must be proved by biopsy) after ASCT, including: Relapse or PD within 12 months after ASCT; if a salvage therapy is received, the patient is non-response (SD or PD) to the last therapy;
6. According to Lugano Criteria (Cheson2014), at least one measurable lesion exists；
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
8. Adequate bone marrow reserve, defined as: Absolute neutrophil count (ANC) ≥1.0×10^9/L; Absolute lymphocyte count (ALC) ≥ 0.3×10^9/L; Platelet (PLT) ≥50×10^9/L;
9. Proper organ function, defined as: Aspartate aminotransferase (AST) ≤ 3 Upper Limit of Normal (ULN); Alanine aminotransferase (ALT) ≤ 3 ULN(AST and ALT≤5 ULN are required for the patients with hepatic dysfunction due to tumor cell infiltration) ; Total serum bilirubin ≤ 2 ULN, unless there exists concurrent Gilbert syndrome; patients with Gilbert syndrome, with total serum bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN, may be included; Serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula); Minimum pulmonary reserve, defined as Grade ≤ 1 dyspnea, and blood oxygen saturation > 91% at non-oxygen inhalation status;
10. Women with child-bearing potential are negative in blood/urine pregnancy tests within 7 d prior to infusion of U16 infusion; any male or female patient with child-bearing potential must agree to adopt effective contraceptive measures throughout the study, and at least one year after administration of the investigational therapy.
11. Qualified T cell function;
12. Vascular conditions for apheresis, and no other contraindications for apheresis;
13. Elution period of CD20 monoclonal antibody at least 3 months before U16 infusion;
14. Life expectancy more than 3 months.

Exclusion Criteria:

1. Patients with other malignant tumors, except for disease-free survival for more than 3 years or carcinoma in-situ;
2. Patients with lymphoma involved with atrium or ventricle；
3. Used immunosuppressants, hormones or high-dose chemotherapy within 2 weeks before signing the informed consent form, or planned to use immunosuppressants or hormones(specifically referring to systemic therapy) before apheresis, except for local or inhaled corticosteroid therapy;
4. Patients complying with any of hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) positive; hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) positive and HBV-DNA copies being more than the lower limit of detection; hepatitis C antibody (HCV-Ab) positive and HBV-RNA copies being more than the lower limit of detection; anti-treponemia pallidum antibody (TP-Ab) positive; Human immunodeficiency virus (HIV) antibody positive; EBV-DNA, and CMV-DNA copies being more than the lower limit of detection;
5. Patients with bacteria, fungi, viruses, mycoplasma or other types of infections, and difficult for controlling by researcher's judgment;
6. Patients with active primary or secondary central nervous system (CNS) lymphoma (a patient with CNS disease symptoms must receive lumbar puncture to exclude CNS lymphoma)；
7. Patients with existing central nervous system disease or with a history of central nervous system disease, e.g., epileptic seizure, cerebral ischemia/hemorrhage, dementia, cerebellum disease, or any autoimmune disease involved with central nervous system；
8. Patients with cardiac angioplasty or stent implantation within 12 months before signing the informed consent form, or myocardial infarction, unstable angina pectoris, other clinically significant heart disease history judged by researcher;
9. Patients need urgent clinical emergencies (such as intestinal obstruction or vascular compression, etc.) due to the obstruction or compression of lymphoma judged by researcher;
10. Patients previously received CAR-T cell therapy with CD20 target;
11. Patients with primary immunodeficiency;
12. Patients who are known with a history of hypersensitivity reaction to any ingredient used for the drug product in the trial.;
13. Patients vaccinated with a live vaccine within 6 weeks prior to screening;
14. Pregnant or lactating women;
15. Patients with active autoimmune diseases;
16. Patients with active acute or chronic graft-versus-host disease (GVHD) when signing the informed consent form;
17. Received allogeneic hematopoietic stem cell transplantation within 6 months before signing the informed consent form;
18. Participated in any other clinical trial within 30 days before signing the i informed consent form;
19. Patients with other conditions that are not suitable to participate in the clinical trial, as considered by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Types, frequency and severity of adverse events | 24 months
  Safty of U16 as measured by types, frequency and severity of adverse events after U16 Injection infusion.
Overall Remission Rate (ORR) | 3 months
  Efficacy of U16 as measured by ORR during the 3 months after U16 Injection infusion, which includes CR and PR.

SECONDARY OUTCOMES:
Complete Remission (CR) | 3 months
  Efficacy of U16 as measured by CR during the 3 months after U16 Injection infusion.
Progression-free survival (PFS) | 24 months
  PFS means duration from the U16 Injection infusion to progression of lymphoma, or death for any reason.
Duration of Remission (DOR) | 24 months
  DOR means the duration from reaching the response (e.g., CR or PR) criteria of the therapy to the first, clearly defined progressive disease, or death for disease under investigation.
Overall Survival（OS） | 24 months
  OS means duration from the U16 Injection infusion to death for any reason, or the last follow-up for survival.
Pharmacokinetic (PK)- Cmax | 24 months
  Maximum detected concentration of U16 in peripheral blood
Pharmacokinetic (PK)- Tmax | 24 months
  Time to maximum concentration of U16 in peripheral blood
Pharmacokinetic (PK)- AUC | 24 months
  Area under the concentration vs time curve of U16 in peripheral blood
Concentration of Cytokines in Serum | 24 months
  Collected as pharmacodynamic data, including IL-6 at least
Concentration of B cells | 24 months
  Measure B cells in peripheral blood

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu